CLINICAL TRIAL: NCT05611931
Title: A Phase 3, Randomized, Placebo-Controlled, Double-Blind, Multicenter Trial of Selinexor in Maintenance Therapy After Systemic Therapy for Patients With p53 Wild-Type, Advanced or Recurrent Endometrial Carcinoma
Brief Title: Selinexor in Maintenance Therapy After Systemic Therapy for Participants With p53 Wild-Type, Advanced or Recurrent Endometrial Carcinoma
Acronym: XPORT-EC-042
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Karyopharm Therapeutics Inc (Industry)
Collaborators: GOG Foundation (Network); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Belgian Gynaecological Oncology Group (Other); North Eastern German Society of Gynaecological Oncology (Other); The Central and Eastern European Gynecologic Oncology Group (Other); Israeli Society of Gynecologic Oncology (Other); Australia New Zealand Gynaecological Oncology Group (Other); Multicenter Italian Trials in Ovarian Cancer (MITO) (Unknown); Grupo Español de Investigación en Cáncer de Ovario (Other); Hellenic Cooperative Oncology Group (HeCOG) (Unknown); Cancer Trials Ireland (CTI) (Unknown); Mario Negri Gynecologic Oncology group (MaNGO) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XPORT-EC-042; GOG-3083 (Other: The GOG Foundation, Inc.); ENGOT-EN20 (Other: European Network of Gynaecological Oncological Trial)
Record Dates: First submitted 2022-11-03; First posted 2022-11-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Endometrial Cancer
Keywords: Selinexor; KPT-330; Advanced or Recurrent Endometrial Carcinoma; XPORT-EC; ENGOT-EN20; GOG-3083; XPORT-EC-042; p53 wild-type; Tumor protein 53 wild-type
MeSH Terms: conditions — Endometrial Neoplasms | interventions — selinexor

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double blind placebo-controlled study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Selinexor (Experimental): Participants will receive a fixed dose of selinexor 60 milligrams (mg) oral tablets once weekly (QW) on Days 1, 8, 15, and 22 of each 28-day cycle.
  Interventions: Drug: Selinexor
- Placebo (Placebo Comparator): Participants will receive matching placebo for selinexor oral tablets QW on Days 1, 8, 15, and 22 of each 28-day cycle.
  Interventions: Drug: Matching Placebo for selinexor

INTERVENTIONS:
Drug: Selinexor — Dose: 60 mg (3 tablets); Dosage form: film-coated, immediate-release tablet of 20 mg each; Route of administration: oral
  Other Names: KPT-330
  Arms: Selinexor
Drug: Matching Placebo for selinexor — Dose:60 mg (3 tablets); Dosage form: film-coated, immediate-release tablet of 20 mg each; Route of administration: oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of selinexor as a maintenance treatment in patients with p53 wt endometrial carcinoma (EC), who have achieved a partial response (PR) or complete response (CR) (per Response Evaluation Criteria in Solid Tumors version 1.1 [RECIST v 1.1]) after completing at least 12 weeks of platinum-based therapy. A total of 276 participants will be enrolled in the study and randomized in a 1:1 ratio to maintenance therapy with either selinexor or placebo.

ELIGIBILITY:
Inclusion Criteria: Patients must meet all of the following inclusion criteria in order to be eligible to participate in this study:

* Adults (Aged ≥ 18 years)
* Histologically confirmed endometrial cancer (endometrioid, serous, undifferentiated, or carcinosarcoma sub-types) that is TP53 wild type by central NGSHistologically confirmed EC including endometrioid, serous, undifferentiated, and carcinosarcoma
* Must have completed at least 12 weeks of platinum-based chemotherapy (with or without immune checkpoint inhibitors), with a confirmed partial or complete response according to RECIST v1.1
* Must be able to initiate C1D1 within 3-8 weeks after last platinum dose
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate bone marrow function and organ function

Exclusion Criteria: Patients meeting any of the following exclusion criteria are not eligible to participate in this study:

* Uterine sarcomas, clear cell or small cell carcinoma with neuroendocrine differentiation
* Palliative radiotherapy administered within 14 days of intended C1D1
* Any gastrointestinal dysfunction that could interfere with the absorption of oral study therapy
* Serious psychiatric or medical conditions that could interfere with study participation or would make study involvement unreasonably hazardous
* Previous treatment with an XPO1 inhibitor
* Stable disease or disease progression after platinum-based chemotherapy
* Pregnancy, breastfeeding, or other legal/ethical restrictions to trial participation
* Known dMMR/MSI-H EC tumors that are medically eligible to receive an immune checkpoint inhibitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 276 (Estimated)
Dates: Start 2023-04-18 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Investigator assessed Progression Free Survival (PFS) per RECIST v1.1 | From randomization until disease progression (PD) or death, whichever occurs first (up to 34 months)

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to 34 months
  Time from randomization to death due to any cause
Safety and tolerability of study drug (selinexor and placebo) | From start of study drug administration up to 34 months
  The safety and tolerability of study drug (selinexor and placebo) will be evaluated based on adverse event (AE) reports, physical examination results (including vital signs), and clinical laboratory results, by means of the occurrence, nature, and severity of AEs via Common Terminology Criteria for Adverse Events (CTCAE) v. 5.0.
Time to First Subsequent Therapy (TFST) | From randomization until date of initiation of first therapy after discontinuation of study drug or death, whichever occurs first (up to 34 months)
  Time from randomization until date of initiation of first therapy after discontinuation of study drug or death, whichever occurs first
Time to Second Subsequent Therapy (TSST) | From randomization until date of initiation of second therapy after discontinuation of study drug or death, whichever occurs first (up to 34 months)
  Time from randomization until date of initiation of second therapy after discontinuation of study drug or death, whichever occurs first
Progression-free survival after initiating a next-line treatment (PFS2) | From randomization until the next-line progression event or death due to any cause, up to 34 months
  Time from randomization until the progression event after initiating a next-line treatment or death due to any cause, whichever occurs first
Progression-free Survival (PFS) as assessed by a Blinded Independent Central Review (BICR), per RECIST v1.1 | From randomization until disease progression (PD) or death, whichever occurs first (up to 34 months)
EuroQol-5 Dimensions-5 Levels Quality of Life Questionnaire (EQ-5D-5L) | From baseline and at specified timepoints up to 34 months
  EQ-5D-5L is a generic questionnaire that assesses health status as perceived by the patient across 5 categories (mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and overall.

CONTACTS AND LOCATIONS:
Locations (217):
- United States (84):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Honor Health, Phoenix, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - UC DAVIS, Davis, California
  - City of Hope National Medical Center, Duarte, California
  - Chao Family Comprehensive Cancer Center and Ambulatory Care, Irvine, California
  - City of Hope at Irvine Lennar, Irvine, California
  - Cancer and Blood Specialty Clinic, Los Alamitos, California
  - UCLA - Women's Health Clinical Research Unit, Los Angeles, California
  - Long Beach Memorial Medical Center, Los Angeles, California
  - UC Irvine, Orange, California
  - Stanford University, Palo Alto, California
  - California Pacific Medical Center, San Francisco, California
  - Highlands Ranch Hospital, Highlands Ranch, Colorado
  - University of Colorado Cancer Center, Highlands Ranch, Colorado
  - Broward Health Medical Center, Fort Lauderdale, Florida
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Advent Health, Orlando, Florida
  - Grady Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Georgia Cancer Center at Augusta University, Augusta, Georgia
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Illinois Cancer Specialists, Arlington Heights, Illinois
  - NorthShore University Health System, Evanston, Illinois
  - Northwest Cancer Center, Dyer, Indiana
  - Goshen Health, Goshen, Indiana
  - St Vincent Hospital, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Iowa, Iowa City, Iowa
  - Our Lady of the Lake Hospital, Inc., Baton Rouge, Louisiana
  - LSU Health Sciences Center New Orleans, New Orleans, Louisiana
  - Trials365, LLC, Shreveport, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - USON - Minnesota Oncology Hematology, Minneapolis, Minnesota
  - University of Minnesota, Minneapolis, Minnesota
  - St. Dominic's Gynecologic Oncology, Jackson, Mississippi
  - Midwest Ventures Group HCA MId America Division, Kansas City, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Intermountain Health St. Vincent Regional Hospital, Billings, Montana
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Center Of Hope, Reno, Nevada
  - Hackensack Meridian Health Jersey Shore University Medical Center, Neptune City, New Jersey
  - Women's Cancer Care Associates, LLC, Albany, New York
  - NYU Langone Hospital-Long Island, Mineola, New York
  - Northwell Health - Zuckerberg Cancer Center, New Hyde Park, New York
  - Mount Sinai Chelsea, New York, New York
  - Perlmutter Cancer Center at NYU Langone Health, New York, New York
  - Mount Sinai, New York, New York
  - Lenox Hill Hospital, New York, New York
  - Northwell Health - Queens Cancer Center, Rego Park, New York
  - University of Rochester, Rochester, New York
  - Atrium Health Levine Cancer Institute, Charlotte, North Carolina
  - Duke Cancer Center, Durham, North Carolina
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - MetroHealth, Cleveland, Ohio
  - Zangmeister Cancer Center, Columbus, Ohio
  - ProMedica Flower Hospital, Sylvania, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute, LLC, Tulsa, Oklahoma
  - Oncology Associates of Oregon, Eugene, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Alliance Cancer Specialists, Langhorne, Pennsylvania
  - Magee - Women's Hospital, Pittsburgh, Pennsylvania
  - Allegheny Health Network - West Penn Hospital, Pittsburgh, Pennsylvania
  - Avera, Sioux Falls, South Dakota
  - Chattanooga's Program in Women's Oncology, Chattanooga, Tennessee
  - The West Clinic, PLLC dba West Cancer Center, Germantown, Tennessee
  - University of Tennessee Medical Center, Knoxville, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - USON - Texas Oncology, Austin Central, Austin, Texas
  - Parkland Health & Hospital System, Dallas, Texas
  - Texas Oncology - Dallas, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Oncology - Fort Worth, Fort Worth, Texas
  - Houston Methodist, Houston, Texas
  - Texas Oncology - San Antonio, San Antonio, Texas
  - Texas Oncology - The Woodlands, The Woodlands, Texas
  - Texas Oncology, PC, Tyler, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Swedish Cancer Institute, Seattle, Washington
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College of Wisconsin/ Freodtert Hospital, Milwaukee, Wisconsin
- Australia (16):
  - Border Medical Oncology & Haematology, Albury, New South Wales
  - Macarthur Cancer Therapy Centre, Campbelltown, New South Wales
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - Central Coast LHD - Gosford & Wyong Hospitals, Gosford, New South Wales
  - Newcastle Private Hospital, New Lambton Heights, New South Wales
  - Royal North Shore Hospital, Saint Leonards, New South Wales
  - Westmead Hospital, Wentworthville, New South Wales
  - ICON Cancer Centre Southport, Southport, Queensland
  - Toowoomba Hospital, Toowoomba, Queensland
  - Royal Hobart Hospital, Hobart, Tasmania
  - Box Hill Hospital - Eastern Health (Oncology), Box Hill, Victoria
  - Monash Health, Clayton, Victoria
  - Frankston Hospital, Frankston, Victoria
  - Cabrini Health, Malvern, Victoria
  - Peter MacCallum Cancer Centre/RWH/RMH, Melbourne, Victoria
  - The Royal Adelaide Hospital, Southport
- Belgium (5):
  - Cliniques Universitaires St. Luc, Brussels
  - AZ Sint Lucas, Ghent
  - UZ Leuven, Leuven
  - CHU Ambroise Pare, Mons
  - CHU UCL Namur, Site Sainte-Elisabeth, Namur
- Canada (8):
  - Tom Baker Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Nova Scotia Health / QEII Health Sciences Centre / Atlantic Clinical Cancer Research Unit, Halifax, Nova Scotia
  - Princess Margaret, Toronto, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Centre Hospitalier de l'Université de Montréal, Montreal, Quebec
  - McGill University Health Centre (MUHC), Montreal, Quebec
  - Hospital Maisonneuve-Rosemont, Montreal, Quebec
- Czechia (5):
  - University Hospital Brno, Brno
  - University Hospital Ostrava, Ostrava
  - UH Královské Vinohrady, Prague
  - General University Hospital in Prague, Prague
  - Hospital Na Bulovce, Prague
- Georgia (8):
  - High Technology Hospital Medcenter, Batumi
  - Todua Clinic, Tbilisi
  - LTD New Hospitals, Tbilisi
  - Tbilisi Cancer Center, Tbilisi
  - JSC - K.Eristavi National Center of Experimental and Clinical Surgery, Tbilisi
  - Caucasus Medical Centre, Tbilisi
  - LTD Innova Medical Center, Tbilisi
  - Multiprofile Clinic "Consilium Medulla", Tbilisi
- Germany (11):
  - Charite Berlin Universitatsmedizin, Berlin
  - Universitätsklinikum Hamburg Eppendorf, Hamburg
  - University Hospital Dresden, Kiel
  - Universitatsklinikum Schleswig-Holstein, Kiel
  - Helios Klinikum Krefeld, Krefeld
  - Universitätsklinik Leipzig, Leipzig
  - Universitätsfrauenklinik Mainz, Mainz
  - Universitätsmedizin Mannheim, Mannheim
  - Klinik und Poliklinik fur Frauenheilkunde und Geburtshilfe GroBhadern, Munich
  - Klinikum Südstadt Rostock, Rostock
  - Universitätsfrauenklinik Ulm, Ulm
- Greece (4):
  - IASO Hospital, Marousi, Athens
  - Alexandra Hospital, Athens
  - Hygeia Hospital, Athens
  - Euromedica General Clinic, Thessaloniki
- Hungary (2):
  - Unit of Gynecol.Oncol., Dept.Obstet.Gynecol., Clinical Center, University of Debrecen, Debrecen
  - Petz Aladár University Teaching Hospital, Győr
- Ireland (5):
  - St. Vincent's University Hospital, Dublin, Elm Park
  - Cork University Hospital, Cork
  - St. James Hospital, Dublin
  - Galway University, Galway
  - University Hospital Waterford, Waterford
- Israel (4):
  - Hillel-Yaffe Medical Center, Hadera
  - Wolfson Medical Center, Holon
  - Hadassah Medical Center, Jerusalem
  - Sheba Medical Center, Ramat Gan
- Italy (15):
  - IRCCS Azienda Ospedaliero Universitaria di Bologna, Bologna
  - ASST Spedali Civili Di Brescia, Brescia
  - IRCCS Istituto Romagnolo Per Lo Studio Del Tumori "Dino Amadori" - IRST S.R.L., Meldola
  - San Raffaele Hospital, Milan
  - Istituto Nazionale dei Tumori IRCCS - MILANO S. C. Ginecologia Oncologica, Milan
  - Instituto Europeo di Oncologia, Milan
  - Humanitas San Pio X Hospital, Milan
  - Ospedale San Gerardo - Asst Monza, Monza
  - "Istituto Nazionale Tumori IRCCS "Fondazione G. Pascale" - NAPOLI Struttura Complessa Oncologia Medica Uro-Ginecologica", Napoli
  - Istituto Oncologico Veneto, Padua
  - Universita di Pisa, Pisa
  - Nuovo Ospedale di Prato, Prato
  - Fondazione Policlinico Universitario Agostino Gemelli - ROMA, Roma
  - Ospedale Ostetrico Ginecologico Sant'Anna, Torino
  - AO Ordine Mauriziano, Torino
- Slovakia (4):
  - St. Elisabeth Cancer Institute, Bratislava
  - UH Bratislava, Bratislava
  - National Cancer Institute, Bratislava
  - UH Trenčín, Trenčín
- South Korea (11):
  - Soon Chun Hyang University Hospital Cheonan, Cheonan, Chungcheongnam-do
  - Severance Hospital (Yonsei University Health System), Seoul, Seongbuk
  - Samsung Changwon Hospital, Changwon
  - National Cancer Center (NCC), Goyang-si
  - CHA University/Bundang CHA General Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Gangnam Severance Hospital, Seoul
  - Seoul National University Bundang Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
- Spain (21):
  - Hospital Universitario Donostia, Donostia / San Sebastian, Gipuzkoa
  - Hospital Clínico Universitario Lozano Blesa, Zaragoza, Zaragoza
  - ICO Badalona, Badalona
  - Hospital Universitari Vall d' Hebrón, Barcelona
  - Hospital Clinic de Barcelona, Barcelona
  - Institut Catala d'Oncologia Hospitalet, Barcelona
  - Hospital Universitario Reina Sofía, Córdoba
  - Institut Catala d'Oncologia de Girona, Girona
  - Hospital Universitario Virgen de las Nieves, Granada
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - Hospital Universitario Clinico San Carlos, Madrid
  - H 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitatrio Virgen de la Victoria, Málaga
  - Virgen de la Arrixaca University Clinical Hospital, Murcia
  - Hospital Universitario Virgen del Rocío, Seville
  - Instituto Valenciano de Oncología, Valencia
  - Hospital Clínico Universitario de Valencia, Valencia
  - Hospital LaFe Uacenlia, Valencia
  - Hospital Miguel Servet, Zaragoza
- Taiwan (7):
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - TaiChung Veterans General Hospital, Taichung
  - Chi Mei Medical Center, Tainan
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Taipei Medical University- Shuang Ho Hospital, Ministry of Health and Welfare, Taipei
  - Chang Gung Memorial Hospital, Taoyuan
- Turkey (Türkiye) (7):
  - Ankara Baskent Hospital, Çankaya, Ankara
  - Çukurova University, Adana
  - Adana Baskent Hospital, Adana
  - Hacettepe University Oncology Hospital, Ankara
  - Memorial Ankara Hospital, Ankara
  - Cerrahpasa University, Istanbul
  - Acibadem Atakent Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Secord AA, Powell MA, McAlpine J. Molecular Characterization and Clinical Implications of Endometrial Cancer. Obstet Gynecol. 2025 Nov 1;146(5):660-671. doi: 10.1097/AOG.0000000000006080. Epub 2025 Sep 18. PMID 40966692
- [Derived] Makker V, Perez-Fidalgo JA, Valabrega G, Hamilton E, Van Gorp T, Sehouli J, Reginacova K, Richardson DL, Perri T, Oza AM, Miller DS, Alia EMG, De Giorgi U, Henry S, Spitz DL, Wimberger P, Bednarikova M, Chon HS, Martinez-Garcia J, Pisano C, Berek JS, Romero I, Scambia G, Farinas-Madrid L, Buscema J, Schochter F, Li K, Kalyanapu P, Walker CJ, Vergote I. Long-term follow-up of efficacy and safety of selinexor maintenance treatment in patients with TP53wt advanced or recurrent endometrial cancer: A subgroup analysis of the ENGOT-EN5/GOG-3055/SIENDO study. Gynecol Oncol. 2024 Jun;185:202-211. doi: 10.1016/j.ygyno.2024.05.016. Epub 2024 Jun 3. PMID 38834399
- [Derived] Vergote I, Perez Fidalgo A, Valabrega G, Monk BJ, Herzog T, Cibula D, Colombo N, Pothuri B, Sehouli J, Korach J, Barlin J, Papadimitriou CA, van Gorp T, Richardson D, McCarthy M, Antill Y, Mirza MR, Li K, Kalyanapu P, Slomovitz B, Coleman RL. ENGOT-EN20/GOG-3083/XPORT-EC-042 - A phase III, randomized, placebo-controlled, double-blind, multicenter trial of selinexor in maintenance therapy after systemic therapy for patients with p53 wild-type, advanced, or recurrent endometrial carcinoma: rationale, methods, and trial design. Int J Gynecol Cancer. 2024 Aug 5;34(8):1283-1289. doi: 10.1136/ijgc-2024-005412. PMID 38627035